CLINICAL TRIAL: NCT00626002
Title: A Phase 3, Multi-center, Open-label Continuation Study in Moderate to Severe Plaque Psoriasis in Subjects Who Completed a Preceding Psoriasis Study With ABT-874
Brief Title: Open Label Continuation Study in Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-016; 2007-005955-40 (EudraCT Number)
Record Dates: First submitted 2008-02-22; First posted 2008-02-29 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Open label
MeSH Terms: interventions — briakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABT-874

INTERVENTIONS:
Drug: ABT-874 — 100mg ABT-874 administered SQ every 4 wks for approximately 204 weeks
  Other Names: briakinumab

SUMMARY:
The purpose of this study is to evaluate long term safety, efficacy and tolerability of ABT-874 in adults with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Having participated in a preceding ABT-874 clinical trial for ABT-874
* Subject has a clinical diagnosis of moderate to severe plaque psoriasis

Exclusion Criteria:

* Subjects who prematurely discontinued in any preceding psoriasis study with ABT-874 other than protocol-required discontinuation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2301 (Actual)
Dates: Start 2008-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving PGA "clear" (0) or "minimal" (1) scores by visit. | Visit (12 weeks)
Proportion of subjects achieving a > PASI 50 clinical response that is defined as a reduction on PASI scores by at least 50% relative to Baseline, by visit. | Visit (12 weeks)
Proportion of subjects achieving a > PASI 75 clinical response that is defined as a reduction on PASI scores by at least 50% relative to Baseline, by visit. | Visit (12 weeks)
AEs, serious adverse events (SAEs), laboratory data, ADA and vital signs will be assessed throughout the study | Visit (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaul, MD, Study Chair — AbbVie
Locations (152):
- United States (98):
  - Site Reference ID/Investigator# 7496, Birmingham, Alabama
  - Site Reference ID/Investigator# 8438, Birmingham, Alabama
  - Site Reference ID/Investigator# 7522, Huntsville, Alabama
  - Site Reference ID/Investigator# 7774, Scottsdale, Arizona
  - Site Reference ID/Investigator# 7435, Tucson, Arizona
  - Site Reference ID/Investigator# 7933, Little Rock, Arkansas
  - Site Reference ID/Investigator# 7234, Bakersfield, California
  - Site Reference ID/Investigator# 8249, Fresno, California
  - Site Reference ID/Investigator# 7332, Irvine, California
  - Site Reference ID/Investigator# 7239, Los Angeles, California
  - Site Reference ID/Investigator# 8390, Oceanside, California
  - Site Reference ID/Investigator# 7503, San Diego, California
  - Site Reference ID/Investigator# 7520, San Diego, California
  - Site Reference ID/Investigator# 7010, San Diego, California
  - Site Reference ID/Investigator# 10962, San Francisco, California
  - Site Reference ID/Investigator# 7334, Santa Monica, California
  - Site Reference ID/Investigator# 7793, Vallejo, California
  - Site Reference ID/Investigator# 7929, Denver, Colorado
  - Site Reference ID/Investigator# 7436, Longmont, Colorado
  - Site Reference ID/Investigator# 7521, New Haven, Connecticut
  - Site Reference ID/Investigator# 7653, Doral, Florida
  - Site Reference ID/Investigator# 8341, Jacksonville, Florida
  - Site Reference ID/Investigator# 7716, Miami, Florida
  - Site Reference ID/Investigator# 7657, Miami, Florida
  - Site Reference ID/Investigator# 10841, South Miami, Florida
  - Site Reference ID/Investigator# 7893, West Palm Beach, Florida
  - Site Reference ID/Investigator# 7331, Alpharetta, Georgia
  - Site Reference ID/Investigator# 9743, Atlanta, Georgia
  - Site Reference ID/Investigator# 7891, Newnan, Georgia
  - Site Reference ID/Investigator# 7932, Snellville, Georgia
  - Site Reference ID/Investigator# 8379, Arlington Heights, Illinois
  - Site Reference ID/Investigator# 8798, Maywood, Illinois
  - Site Reference ID/Investigator# 10703, Schaumburg, Illinois
  - Site Reference ID/Investigator# 6950, Skokie, Illinois
  - Site Reference ID/Investigator# 7892, West Dundee, Illinois
  - Site Reference ID/Investigator# 6933, Indianapolis, Indiana
  - Site Reference ID/Investigator# 10422, Indianapolis, Indiana
  - Site Reference ID/Investigator# 16581, Plainfield, Indiana
  - Site Reference ID/Investigator# 7992, Overland Park, Kansas
  - Site Reference ID/Investigator# 17193, Henderson, Kentucky
  - Site Reference ID/Investigator# 8528, Louisville, Kentucky
  - Site Reference ID/Investigator# 9962, Owensboro, Kentucky
  - Site Reference ID/Investigator# 8529, Andover, Massachusetts
  - Site Reference ID/Investigator# 8149, Boston, Massachusetts
  - Site Reference ID/Investigator# 9823, Detroit, Michigan
  - Site Reference ID/Investigator# 7883, Fort Gratiot, Michigan
  - Site Reference ID/Investigator# 7238, Grand Blanc, Michigan
  - Site Reference ID/Investigator# 7656, Fridley, Minnesota
  - Site Reference ID/Investigator# 6930, St Louis, Missouri
  - Site Reference ID/Investigator# 6949, St Louis, Missouri
  - Site Reference ID/Investigator# 7240, Omaha, Nebraska
  - Site Reference ID/Investigator# 9567, Omaha, Nebraska
  - Site Reference ID/Investigator# 7757, Berlin, New Jersey
  - Site Reference ID/Investigator# 7330, East Windsor, New Jersey
  - Site Reference ID/Investigator# 7882, New Brunswick, New Jersey
  - Site Reference ID/Investigator# 7455, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 8078, Buffalo, New York
  - Site Reference ID/Investigator# 8392, New York, New York
  - Site Reference ID/Investigator# 8006, New York, New York
  - Site Reference ID/Investigator# 7230, New York, New York
  - Site Reference ID/Investigator# 10201, New York, New York
  - Site Reference ID/Investigator# 8037, Rochester, New York
  - Site Reference ID/Investigator# 7333, Stoney Brook, New York
  - Site Reference ID/Investigator# 7434, Hickory, North Carolina
  - Site Reference ID/Investigator# 8117, Wilmington, North Carolina
  - Site Reference ID/Investigator# 9681, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 6945, Cincinnati, Ohio
  - Site Reference ID/Investigator# 23345, Cincinnati, Ohio
  - Site Reference ID/Investigator# 7044, Cleveland, Ohio
  - Site Reference ID/Investigator# 7899, Columbus, Ohio
  - Site Reference ID/Investigator# 8389, Dayton, Ohio
  - Site Reference ID/Investigator# 11181, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 6936, Lake Oswego, Oregon
  - Site Reference ID/Investigator# 7703, Portland, Oregon
  - Site Reference ID/Investigator# 6948, Portland, Oregon
  - Site Reference ID/Investigator# 11424, Portland, Oregon
  - Site Reference ID/Investigator# 8494, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 7930, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 6934, Johnston, Rhode Island
  - Site Reference ID/Investigator# 6935, Providence, Rhode Island
  - Site Reference ID/Investigator# 7785, Greer, South Carolina
  - Site Reference ID/Investigator# 7497, Goodlettsville, Tennessee
  - Site Reference ID/Investigator# 7388, Knoxville, Tennessee
  - Site Reference ID/Investigator# 6931, Nashville, Tennessee
  - Site Reference ID/Investigator# 7684, Arlington, Texas
  - Site Reference ID/Investigator# 10842, Austin, Texas
  - Site Reference ID/Investigator# 7498, Dallas, Texas
  - Site Reference ID/Investigator# 6947, Dallas, Texas
  - Site Reference ID/Investigator# 6944, Houston, Texas
  - Site Reference ID/Investigator# 7758, San Antonio, Texas
  - Site Reference ID/Investigator# 8108, San Antonio, Texas
  - Site Reference ID/Investigator# 6937, Tyler, Texas
  - Site Reference ID/Investigator# 7655, Webster, Texas
  - Site Reference ID/Investigator# 10207, Salt Lake City, Utah
  - Site Reference ID/Investigator# 6946, Norfolk, Virginia
  - Site Reference ID/Investigator# 6932, Seattle, Washington
  - Site Reference ID/Investigator# 10306, Spokane, Washington
  - Site Reference ID/Investigator# 7884, Milwaukee, Wisconsin
- Austria (2):
  - Site Reference ID/Investigator# 16845, Graz
  - Site Reference ID/Investigator# 18183, Vienna
- Site Reference ID/Investigator# 15761, Brussels, Belgium
- Canada (23):
  - Site Reference ID/Investigator# 7991, Barrie
  - Site Reference ID/Investigator# 8047, Calgary
  - Site Reference ID/Investigator# 7996, Edmonton
  - Site Reference ID/Investigator# 6996, Halifax
  - Site Reference ID/Investigator# 7236, Hamilton
  - Site Reference ID/Investigator# 6995, Laval
  - Site Reference ID/Investigator# 6998, London
  - Site Reference ID/Investigator# 7043, London
  - Site Reference ID/Investigator# 7329, Markham
  - Site Reference ID/Investigator# 6999, Montreal
  - Site Reference ID/Investigator# 7652, Montreal
  - Site Reference ID/Investigator# 7006, North Bay
  - Site Reference ID/Investigator# 8102, Ottawa
  - Site Reference ID/Investigator# 6993, Québec
  - Site Reference ID/Investigator# 8112, St. John's
  - Site Reference ID/Investigator# 7931, Surrey
  - Site Reference ID/Investigator# 8118, Vancouver
  - Site Reference ID/Investigator# 6997, Vancouver
  - Site Reference ID/Investigator# 6994, Waterloo
  - Site Reference ID/Investigator# 8111, Westmount
  - Site Reference ID/Investigator# 7005, Windsor
  - Site Reference ID/Investigator# 7979, Windsor
  - Site Reference ID/Investigator# 8348, Winnipeg
- Denmark (2):
  - Site Reference ID/Investigator# 17781, Aarhus
  - Site Reference ID/Investigator# 18041, Copenhagen NV
- Finland (4):
  - Site Reference ID/Investigator# 18661, Helsinki
  - Site Reference ID/Investigator# 18701, Kuopio
  - Site Reference ID/Investigator# 14962, Lahti
  - Site Reference ID/Investigator# 19241, Turku
- France (3):
  - Site Reference ID/Investigator# 18502, Nice
  - Site Reference ID/Investigator# 16781, Paris
  - Site Reference ID/Investigator# 18506, Toulouse
- Germany (7):
  - Site Reference ID/Investigator# 16281, Berlin
  - Site Reference ID/Investigator# 15664, Frankfurt am Main
  - Site Reference ID/Investigator# 15663, Hamburg
  - Site Reference ID/Investigator# 16381, Kiel
  - Site Reference ID/Investigator# 16143, Munich
  - Site Reference ID/Investigator# 16161, Münster
  - Site Reference ID/Investigator# 17676, Tübingen
- Greece (3):
  - Site Reference ID/Investigator# 16282, Athens
  - Site Reference ID/Investigator# 15921, Athens
  - Site Reference ID/Investigator# 15922, Thessaloniki
- Italy (2):
  - Site Reference ID/Investigator# 15401, Modena
  - Site Reference ID/Investigator# 14881, Rome
- Spain (2):
  - Site Reference ID/Investigator# 19322, Barcelona
  - Site Reference ID/Investigator# 15341, Madrid
- Site Reference ID/Investigator# 16142, Stockholm, Sweden
- Switzerland (2):
  - Site Reference ID/Investigator# 17721, Geneva
  - Site Reference ID/Investigator# 16749, Zurich
- United Kingdom (2):
  - Site Reference ID/Investigator# 19045, Aberdeen
  - Site Reference ID/Investigator# 15422, Manchester